CLINICAL TRIAL: NCT00544856
Title: Effects of a Complex Cognitive Training in Mild Cognitive Impairment and Mild Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: cogT001
Record Dates: First submitted 2007-10-12; First posted 2007-10-16 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Alzheimer's Disease; Cognitive Impairment
Keywords: mild Alzheimer's disease; mild cognitive impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental): cognitive intervention
  Interventions: Behavioral: complex cognitive training
- 2 (Placebo Comparator)
  Interventions: Behavioral: complex cognitive training

INTERVENTIONS:
Behavioral: complex cognitive training

SUMMARY:
A recent meta-analysis that included over 29.000 individuals found that the odds ratio (OR) of individuals with high brain reserve compared to low was 0.54 (p < 0.0001), a risk decrease of 46%. Among the factors that influence cognitive reserve, mentally stimulating activities was the most robust factor after controlling for education, age, occupation and other potential confounds. The brain reserve effect was sustained over a median longitudinal follow-up of 7 years. It would be interesting to detect whether a complex cognitive training could show similar effects on the cognitive abilities of patients with mild Alzheimer's disease (AD) and mild cognitive impairment (MCI) as it has been reported in previous studies based on mentally stimulating activities analysis.

The hypothesis is that a complex cognitive training alters the neural networks in both subject groups and this alteration is associated with improvement or stabilization of cognitive and non-cognitive function.

The investigator will perform a complex cognitive training program. Twenty patients with mild AD and twenty four patients with MCI will be recruited in this study. The patients will be randomised in control- and treatment groups.Additionally indirect effects on non-cognitive functions will be evaluated in caregivers of the patients.

The investigators expect that the cognitive and non-cognitive abilities will be changed during the cognitive training. The investigators also expect differences between treatment and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 55 years, fulfilling criteria of the National Institute of Neurological and Communicative Disease and Stroke (NINCDS) and the Alzheimer's Disease and Related Disorders Association (ADRDA) for the diagnosis of clinically probable AD or Petersen's criteria of mild cognitive impairment (MCI)
* No evidence for other psychiatric axis I disorders according to DSM-IV criteria
* No uncontrolled arterial hypertension or diabetes mellitus
* No history of drug/alcohol abuse
* Cholinesterase inhibitors or Memantine must have been in a stabile doses at least 2 moths in AD subject group prior to the Baseline
* The patient is able to provide written informed consent to participate in the study. If, at investigator's discretion, a patient is considered not to be capable to give legal consent, then written consent must also be obtained from the patient's legally acceptable representative.

Exclusion Criteria:

* Evidence for other psychiatric axis I disorders according to DSM-IV criteria
* Uncontrolled arterial hypertension or diabetes mellitus
* History of drug/alcohol abuse
* No ability to participate and no willing to give informed consent and comply with the study restrictions

Ages: 55 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 39
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
cognition: MMSE, ADAS-cog. | month 0, 6, 12

SECONDARY OUTCOMES:
quality of life | month 0, 6, 12

CONTACTS AND LOCATIONS:
Overall Officials: Harald Hampel, MD, Study Chair — Department of Psychiatry, Ludwig-Maximilian University, Munich Germany

REFERENCES:
- [Derived] Buschert VC, Giegling I, Teipel SJ, Jolk S, Hampel H, Rujescu D, Buerger K. Long-term observation of a multicomponent cognitive intervention in mild cognitive impairment. J Clin Psychiatry. 2012 Dec;73(12):e1492-8. doi: 10.4088/JCP.11m07270. PMID 23290333